CLINICAL TRIAL: NCT06660914
Title: A Randomized Controlled Trial Comparing Robotic Flexible Ureteroscopy With Standard Flexible Ureteroscopy for Treatment of Renal Stones - A Pilot Study
Brief Title: Robotic Flexible Ureteroscopy Versus Standard Flexible Ureteroscopy for Renal Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE-2024.217
Record Dates: First submitted 2024-10-14; First posted 2024-10-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic flexible ureteroscopy with ILY® Robot platform (Experimental): Robotic ILY® is a flexible ureteroscopy holder with multiple degrees of freedom telemanipulated with a wireless controller. This allows the surgeon to work easily at a distance from the patient and prevents them from exposing to the source of ionizing radiation.
  Interventions: Procedure: Flexible Ureteroscopy
- Standard flexible ureteroscopy (Active Comparator): Standard flexible ureterscopy
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Flexible Ureteroscopy — Ureteroscopic lithotripsy

SUMMARY:
This is a prospective randomized clinical trial which aims to compare the clinical outcomes of robotic flexible ureteroscopy and standard flexible ureteroscopy for the treatment of renal stones.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial comparing robotic flexible ureteroscopy and standard flexible ureteroscopy for patients with treatment of renal stones. All consecutive patients who are scheduled for flexible ureteroscopy for treatment of renal stones would be screened for study eligibility. Patients are randomised to receive either robotic or standard flexible ureteroscopy with an allocation ratio of 1:1. by computer generated random block. The urologist performing the surgery could not be blinded due to the nature of the intervention. Patients receiving the treatment and investigators assessing for any disease recurrence are blinded from the allocated treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old with informed consent
* Being willing and able to provide written informed consent

Exclusion Criteria:

* Patients with abnormal urinary tract (e.g. ileal conduit, neobladder, ureteric stricture)
* American Society of Anesthesiologists (ASA) physical status classification system >3
* Untreated urinary tract infection
* Renal stones > 3cm in diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate at 1 month | Month 1
  Stone-free rate at 1 month is defined by non contrast computer tomography (NCCT) performed within 24 hours of surgery without residual stone fragments or residual stone fragments <2mm

SECONDARY OUTCOMES:
Stone-free rate at 3 month | Month 3
  If not stone free at 1 month, stone-free rate at 3 month is defined by non contrast computer tomography (NCCT) performed within 24 hours of surgery without residual stone fragments or residual stone fragments <2mm
Operative time | During operation
  the time from insertion of an endoscope into the urethra to the completion of stent placement
Lasing Time | During operation
  The total lasing time in minutes during operation
Total laser energy used | During operation
  Total laser energy used during operation
Total radiation dose | During operation
  Total radiation dose during operation
Total radiation time | during operation
  total radiation time in minutes during operation
Length of hospital stay | On Discharge
  defined from the day of surgery to the day of discharge, counted in days.
Postoperative pain | Baseline, Week 1 and Week 12
  By visual analogue scores from 0-10, the highest score the more pain.
Surgeon radiation exposure | During operation
  By radiation dosimeter

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- North District Hospital, Sheung Shui, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bravo-Balado A, Fontanet S, Skolarikos A, Gozen AS, Somani BK, Traxer O, Papatsoris A, Ruiz Martinez A, Keller EX, Pietropaolo A, Tonyali S, Tailly T, Esperto F, Liatsikos E, Kanashiro AK, Angerri O, Emiliani E. Estimated Radiation Dose to the Lens During Endourologic Procedures: The Role of Leaded Glasses and the ALARA Protocol-An ESU/ESUT-YAU Endourology Group Collaboration. J Endourol. 2023 Aug;37(8):935-939. doi: 10.1089/end.2023.0061. PMID 37337653
- [Background] Desai MM, Grover R, Aron M, Ganpule A, Joshi SS, Desai MR, Gill IS. Robotic flexible ureteroscopy for renal calculi: initial clinical experience. J Urol. 2011 Aug;186(2):563-8. doi: 10.1016/j.juro.2011.03.128. Epub 2011 Jun 16. PMID 21683380
- [Background] Geavlete P, Saglam R, Georgescu D, Multescu R, Iordache V, Kabakci AS, Ene C, Geavlete B; -. Robotic Flexible Ureteroscopy Versus Classic Flexible Ureteroscopy in Renal Stones: the Initial Romanian Experience. Chirurgia (Bucur). 2016 Jul-Aug;111(4):326-9. PMID 27604670
- [Background] El-Hajj A, Abou Chawareb E, Zein M, Wahoud N. First prospective clinical assessment of the ILY(R) robotic flexible ureteroscopy platform. World J Urol. 2024 Mar 13;42(1):143. doi: 10.1007/s00345-024-04869-7. PMID 38478076
- [Background] Klein J, Charalampogiannis N, Fiedler M, Wakileh G, Gozen A, Rassweiler J. Analysis of performance factors in 240 consecutive cases of robot-assisted flexible ureteroscopic stone treatment. J Robot Surg. 2021 Apr;15(2):265-274. doi: 10.1007/s11701-020-01103-5. Epub 2020 Jun 16. PMID 32557097
- [Background] Tae BS, Balpukov U, Cho SY, Jeong CW. Eleven-year Cumulative Incidence and Estimated Lifetime Prevalence of Urolithiasis in Korea: a National Health Insurance Service-National Sample Cohort Based Study. J Korean Med Sci. 2018 Jan 8;33(2):e13. doi: 10.3346/jkms.2018.33.e13. PMID 29215822
- [Background] Sorokin I, Mamoulakis C, Miyazawa K, Rodgers A, Talati J, Lotan Y. Epidemiology of stone disease across the world. World J Urol. 2017 Sep;35(9):1301-1320. doi: 10.1007/s00345-017-2008-6. Epub 2017 Feb 17. PMID 28213860
- [Background] Geraghty R, Abourmarzouk O, Rai B, Biyani CS, Rukin NJ, Somani BK. Evidence for Ureterorenoscopy and Laser Fragmentation (URSL) for Large Renal Stones in the Modern Era. Curr Urol Rep. 2015 Aug;16(8):54. doi: 10.1007/s11934-015-0529-3. PMID 26077357
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Park IW, Kim SJ, Shin D, Shim SR, Chang HK, Kim CH. Radiation exposure to the urology surgeon during retrograde intrarenal surgery. PLoS One. 2021 Mar 15;16(3):e0247833. doi: 10.1371/journal.pone.0247833. eCollection 2021. PMID 33720938
- [Background] Mansoor SN, Al Arabia DH, Rathore FA. Ergonomics and musculoskeletal disorders among health care professionals: Prevention is better than cure. J Pak Med Assoc. 2022 Jun;72(6):1243-1245. doi: 10.47391/JPMA.22-76. PMID 35751350
- [Background] Allaire PE, Kim HC, Maslen EH, Olsen DB, Bearnson GB. Prototype continuous flow ventricular assist device supported on magnetic bearings. Artif Organs. 1996 Jun;20(6):582-90. PMID 8817961